CLINICAL TRIAL: NCT03919110
Title: Immunome Project Consortium for Autoinflammatory Disorders
Acronym: ImmunAID
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C18-30
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2023-11

CONDITIONS: Autoinflammatory Diseases, Hereditary
Keywords: Inflammation; Rheumatology
MeSH Terms: conditions — Hereditary Autoinflammatory Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, cells, DNA, as well as urine and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Genetically Undiagnosed SAID Patients (guSAID): adults and children, with different SAID of unknown pathogenesis, for which no specific mutations is identified and whose pathogenic mechanism remains unknown:
  * Still Disease,
  * Recurrent pericarditis,
  * Neutrophilic dermatosis,
  * Schnitzler,
  * Vasculitis (Kawasaki disease, Behçet disease, Takayasu arteritis),
  * Inflammation of unknown origin,
  * Chronic/recurrent osteitis.
  Interventions: Diagnostic Test: Collection of biological samples
- Parents of guSAID patients: Enrollment of parents of guSAID patients is justified by the TRIO genomic analysis (patient plus two parents) of the guSAID patients without known mutations. Indeed, the TRIO based whole-exome sequencing helps to facilitate the interpretation of genotypes and improve genetic explorations
  Interventions: Diagnostic Test: Collection of biological samples
- Monogenic SAID patients (mSAID): This group of patients will serve as positive control to classify other diseases and encompass the following diseases: FMF, TRAPS, HIDS, and CAPS. Investigators aim at recruiting 50 patients per disease entity.
  Interventions: Diagnostic Test: Collection of biological samples
- Patient Free of inflammatory disorders control subjects: In order to set a reference / baseline for the identification of biomarkers the study will need non-inflammatory samples.
  Interventions: Diagnostic Test: Collection of biological samples

INTERVENTIONS:
Diagnostic Test: Collection of biological samples — Investigators are building a collection of biological samples to perform biological assays and multiple analyses so-called "omics": genomics (on the entire genome), proteomics (on all proteins) etc...This will make it possible to identify the genetic mutations or biological markers present or absent in these diseases, making it possible to confirm a diagnosis or to eliminate differential diagnoses.

SUMMARY:
Rare systemic auto inflammatory diseases are a group of diseases that can be inherited and have non specific symptoms (fevers, rashes, joint pain, etc.). These diseases can be divided into two groups:

* Diseases for which genetic mutations have been identified
* The so-called genetically undetermined diseases for which no genetic mutation has been identified and for which the diagnosis is based on the elimination of other causes of disease

At present, the causes and mechanisms of these diseases are poorly understood and their diagnosis is difficult, often leading to misdiagnosis. The usual care integrates anti-inflammatory treatments (aspirin, colchicine, cortisone, biotherapies, etc.) and support for patients and their families by health professionals (doctors, nurses, physiotherapists, etc.). To date, a patient with one of these diseases can receive up to 5 inappropriate or ineffective treatments before the right diagnosis is made and the right therapy is put in place.

The objective of this study is to develop rapid and effective diagnostic methods for these diseases by the identification of biological markers present in blood, urine or stool of patient in order to develop a rapid and efficient diagnostic method.

DETAILED DESCRIPTION:
The objective of this study is to develop rapid and effective diagnostic methods for these diseases by the identification of biological markers present in blood, urine or stool of patient in order to develop a rapid and efficient diagnostic method. To this end, investigators are building a collection of biological samples derived from blood (plasma, serum, cells and DNA) as well as urine and stool to perform biological assays and multiple analyses so-called "omics": genomics (on the entire genome), proteomics (on all proteins) etc...This will make it possible to identify the genetic mutations or biological markers present or absent in these diseases, making it possible to confirm a diagnosis or to eliminate differential diagnoses.

To better understand and identify the abnormalities leading to the onset of auto-inflammatory diseases, four groups will be constituted:

* a group of patients with auto-inflammatory diseases for which a genetic mutation has been identified.
* a group of subjects free from any auto-inflammatory disease.
* a group of patients suffering from an auto-inflammatory disease, poorly characterized; i.e. auto-inflammatory diseases for which clinicians are not certain on mechanisms leading to the onset of the disease.
* a group of parents of patients suffering from an auto-inflammatory disease, poorly characterized.

At a routine follow-up visit, the investigator will inform the participant about the nature and purpose of the study research.

If the participant agree, the participant will sign the consent to participate in this study and the tests investigators will administer for this study will take place during a consultation of approximately 2 hours.

In order to carry out the biological assays as well as the multiple "omics" analyses (genomics (on the whole genome), proteomics (on all proteins)), a blood sample will be taken depending on your weight and age and according to the recommendation in force (maximum of 11 × 7 mL).

The participant will also be asked to collect urine and stool using a kit designed for this purpose.

This research requires collecting from participant medical file the personal demographic data, medical data, medical imaging results and biological and genetic analyses. All these analyses will have been carried out as part of the diagnosis and management of participant disease.

Investigators will collect participant laboratory test results (immunology, serology, biochemistry, genetics...) in order to describe the characteristics of their disease.

During patient participation and in order to assess your quality of life, particiapnts will be asked to complete a specific questionnaire (SF-36, about 15 minutes). During this consultation you will also be asked to complete (i) a simple questionnaire that describes your functional abilities (HAQ, about 10 minutes), (ii) the AIDAI (Auto-inflammatory Disease Activity Index) score that allows you to evaluate the activity of your auto-inflammatory disease and (iii) a questionnaire focusing on your diet and gut function.

Depending on the case, a follow-up consultation at 3 months may be offered by the investigator. This visit will last a maximum of one hour and will be combined with a new blood test, a urine and stool collection and the completion of a questionnaire on diet and gut function .

Finally, a 12-month follow-up survey may be conducted by the investigator (by telephone or by medical file) to ensure your health status, for the sole purpose of the research.

ELIGIBILITY:
Inclusion Criteria for guSAID Patients

* SAID patients with an as yet unidentified genetic cause.
* Patients diagnosed according to the specific diagnostic criteria of each diseases. For each - subgroup, the diagnosis will be based on accepted criteria.
* Patients with active disease (presence of a flare) according to the specific criteria for each disease (Cf. Table 2)
* For age criteria, please refer to each subgroup
* Patients covered by a health insurance
* Signature of the informed consent (parents/legal representative if the patient is less than <18 years old)

Exclusion Criteria for guSAID Patients:

* Active chronic infection included chronic viral infection (HIV, HBV, HCV…)
* Recent infection or antibiotic treatment in the last 2 weeks
* Systemic auto-immune disease
* Other etiology of fever (infection or neoplasia)
* Monogenic auto-inflammatory disease (other than FMF, HIDS, TRAPS, CAPS)
* Genetic macrophage activation syndrome
* Evidence of immuno-deficiency (e.g., transplant recipient, immunosuppressive treatment for other conditions etc.)
* Pregnancy
* Individuals deprived of liberty
* Inability to understand the local language
* Protected persons (under guardianship or curatorship)

Inclusion criteria for parents of guSAID patients

* First-degree biological relationship (no adoption) with the index patient
* Mother and Father aged more than 18 years old
* Health insurance coverage
* Signature of the informed consent form

Exclusion criteria for parents of guSAID patients

* Any condition which in the Investigator's opinion makes it undesirable for the subject to -
* participate in the study or which would jeopardize compliance with the protocol
* Individuals deprived of liberty
* Inability to understand the local language
* Protected persons

Inclusion criteria for mSAID patients

* Patients with monogenic hereditary SAID
* Patients diagnosed according to the specific diagnostic criteria of each diseases. EUROFEVER criteria for clinical definition plus genetic criterion
* Patients with active disease (presence of a flare and/ or persistent chronic inflammation) :
* Patients older than 6 months can be recruited
* Patients with health insurance
* Signature of the informed consent form

Exclusion criteria for mSAID Patients

* Active chronic infection included chronic viral infection (HIV, HBV, HCV…)
* Recent infection or antibiotic treatment
* Systemic auto-immune disease
* Other etiology of fever (infection or neoplasia)
* Monogenic auto-inflammatory disease (other than FMF, HIDS, TRAPS, CAPS)
* Genetic macrophage activation syndrome
* Evidence of immuno-deficiency
* Pregnancy
* Individuals deprived of liberty
* Inability to understand the local language
* Protected persons

Inclusion criteria for negative control

* Subject free of inflammatory disorders and negative CRP at enrollment
* Subject without personal or familial history of SAID
* Subject aged from 10 to 60 years old
* Subject with health insurance
* Signature of the informed consent form

Exclusion criteria for negative control

* Active bacterial, viral, fungal, or opportunistic infections
* Recent infection or antibiotic treatment in the last 2 weeks
* History of any inflammatory, auto-inflammatory or auto-immune disease
* History of systemic corticosteroid or non-steroidal (NSAID) therapy within the last 4 weeks
* History of neoplasia with the exception of adequately treated basal and squamous cell -
* carcinoma of the skin, or carcinoma in situ of the cervix
* Evidence of immunocompromised
* End stage renal disease (eGFR <20 mL/min/1.73m2)
* Comorbidities requiring corticosteroid therapy, including those which have required three or more courses of systemic corticosteroids within the previous 12 months
* Pregnancy
* Current substance abuse or history of substance abuse within the past year.
* Lack of peripheral venous access
* Individuals deprived of liberty
* Inability to understand the local language
* Protected persons (under guardianship or curatorship)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1616 subjects will be recruited. Four groups will be constituted:
  * patients with auto-inflammatory diseases for which a genetic mutation has been identified. This population will be the positive control.
  * subjects free from any auto-inflammatory disease. It will be the negative control.
  * patients suffering from an auto-inflammatory disease, poorly characterized;
  * parents of patients suffering from an auto-inflammatory disease, poorly characterized.
Sampling Method: Non-Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | [0-6] MONTHS
  Area under the curve (AUC) of the candidate algorithm able to discriminate between healthy controls and patients with SAID, either monogenic SAIDs (positive controls) or undiagnosed SAIDs.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FAUTREL, MD, PhD, Principal Investigator — Department of RHeumatology, Groupe Hospitalier Pitié-Salpêtrière; Christian von FRENCKELL, MD, PhD, Principal Investigator — CHU de Liège, Department of Rheumatology; Vassili SOUMELIS, MD,PhD, Study Director — INSERM U932
Locations (1):
- Hôpital Universitaire Pitié Salpêtrière, Paris, France